CLINICAL TRIAL: NCT06925529
Title: Protecting Neurovascular Function In lOng-term Breast caNcer Survivors With ExercisE tRaining - The PIONEER Study
Brief Title: Exercise to Improve Neurovascular Function in Breast Cancer Survivors
Acronym: PIONEER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P11723; 114949 (Other: Alfred HREC)
Record Dates: First submitted 2025-03-20; First posted 2025-04-13 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Survivorship
Keywords: Breast Cancer; Survivorship; Neurovascular Function; Cerebral Blood Flow; Cardio-Oncology; Exercise Training; Neurocognitive Function
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care (No Intervention): Participants randomised to the usual care group will be provided with their usual care by their usual healthcare professional(s). The usual care group will not be prescribed any exercise training through the study. However, they will be informed that they should aim to achieve the physical activity and exercise guidelines for Australian adults or older adults depending on their age (Care, 2024). The usual care group will not be monitored throughout the study intervention period, except for the reporting of adverse events where necessary.
- Cardio-Oncology Rehabilitation and Exercise Programme (Experimental): Participants randomised to the CORE programme will receive exercise training that is analogous to cardiac rehabilitation, but Exercise Physiologists will individualise each training program using the participants baseline CPET results to maximise adherence and improve the effectiveness of the training program beyond typical cardiac rehabilitation programs. An Exercise Physiologist will supervise two training sessions a week and monitor adherence to one other independent session at home each week for the first 12 weeks of the training program whilst exercise frequency, intensity, and time is progressively increased. Supervision of the exercise training will then be stepped down gradually after 12 weeks to a fortnightly check-in to encourage intervention adherence. Patients will be provided with a training calendar and objective tools for tracking physical activity (e.g. heart rate monitor and diary). Adherence will be monitored in real-time using a research web-based platform.
  Interventions: Behavioral: Cardio-Oncology Rehabilitation and Exercise Programme

INTERVENTIONS:
Behavioral: Cardio-Oncology Rehabilitation and Exercise Programme — Participants randomised to the CORE programme will receive exercise training that is analogous to cardiac rehabilitation, but Exercise Physiologists will individualise each training program using the participants baseline CPET results to maximise adherence and improve the effectiveness of the training program beyond typical cardiac rehabilitation programs. An Exercise Physiologist will supervise two training sessions a week and monitor adherence to one other independent session at home each week for the first 12 weeks of the training program whilst exercise frequency, intensity, and time is progressively increased. Supervision of the exercise training will then be stepped down gradually after 12 weeks to a fortnightly check-in to encourage intervention adherence. Patients will be provided with a training calendar and objective tools for tracking physical activity (e.g. heart rate monitor and diary). Adherence will be monitored in real-time using a research web-based platform.
  Other Names: Exercise Training
  Arms: Cardio-Oncology Rehabilitation and Exercise Programme

SUMMARY:
Study Rationale:

Breast cancer survivors are more likely to develop cardiovascular disease (CVD) or neurocognitive disease than age-matched counterparts without a history of cancer diagnosis. Some anti-cancer treatments cause damage to the cells of heart and the walls of blood vessels, which may exacerbate neurovascular dysfunction and cancer-related cognitive impairment (symptoms such as 'chemo-brain'), as well as accelerating the onset of neurocognitive disease. Therefore, effective policies and therapeutic strategies are needed to minimize neurovascular dysfunction and neurocognitive disease in at-risk populations like breast cancer survivors.

Regular exercise training is effective in slowing or preventing the development of CVD. Furthermore, higher fitness levels are associated with lower dementia risk in older adults, which may be due to better neurovascular function. However, whether exercise training incorporated into a Cardio-Oncology Rehabilitation and Exercise (CORE) programme can improve neurovascular function in breast cancer survivors is currently unknown. Therefore, the primary aim of this study will be to determine the effect of a CORE programme on neurovascular function in long-term breast cancer survivors.

Study Description:

This study will be a randomised controlled trial to investigate the effect of a CORE programme on neurovascular function in long-term breast cancer survivors.

Participants will complete a series of baseline assessments, including lifestyle questionnaires, a cognitive function assessment, dual-energy x-ray absorptiometry (DXA), a cardiopulmonary exercise test (CPET), ultrasound assessments of arterial stiffness and vascular function, and brain magnetic resonance imaging (MRI). Furthermore, participants will wear a blood pressure monitor at home for 24 hours, and a physical activity monitor for seven days.

Following completion of baseline assessments, participants will be randomised to either the CORE program or a 'usual care' group. The CORE program will include a 6-month exercise training program supervised by an Exercise Physiologist at the Baker Heart and Diabetes Institute. The usual care group will carry on with healthcare from their usual healthcare provider(s) for 6 months.

Participants will then complete two follow-up study visits following completion of the 6-month intervention period, with identical procedures to the baseline study visits.

Study Duration:

This study involves two baseline study visits in month 1, followed by two study visits in month 7. Participants randomised to the CORE program will be asked to attend the Baker Heart and Diabetes Institute on a weekly basis for supervised exercise training sessions. However, the supervised exercise training sessions will be provided by a mix of in-person, video-conferencing and tele-health modes depending on each participants availability and needs.

DETAILED DESCRIPTION:
Study Rationale:

Breast cancer (BC) is the most common diagnosed cancer in Australian females (BreastScreen Australia Monitoring Report 2024, Summary, 2024). Although the 5-year relative survival from a stage 1 - 3 BC diagnosis is improving due to earlier screening and more targeted treatment plans (Breast Cancer in Australia, 2012), females with a previous BC diagnosis are more likely to develop cardiovascular disease (CVD) or neurocognitive disease than age-matched counterparts without a previous BC diagnosis (Lange et al., 2019).

Aging is a major risk factor for CVD (Deaths in Australia, Leading Causes of Death, 2024) and neurocognitive disease (Dementia in Australia, Summary, 2024). Australians over the age of 65 years old currently account for 16% of the population, but this is expected to increase to 23% by 2066 (Older Australians, Demographic Profile - Australian Institute of Health and Welfare, 2024). Furthermore, the majority (69%) of BC cases are diagnosed in females aged 40-69 (Breast Cancer in Australia, 2012). As such, the number of females diagnosed with BC is expected to increase given the ageing population, and a as result, so too will the number of long-term BC survivors diagnosed with either CVD, neurocognitive disease, or both. Therefore, effective policies and therapeutic strategies are needed to minimize the growing societal and economic burden of CVD and neurocognitive disease, with particular focus on high-risk populations like BC survivors.

The clustering of CVD risk factors and the cardiotoxic effects of anti-cancer treatments (e.g. anthracycline-based chemotherapy and radiotherapy to the left side of the chest) contribute to the higher prevalence of CVD in BC survivors (Yeh & Bickford, 2009). While the exact mechanisms are currently unclear, the increasing burden of neurocognitive disease and cancer-related cognitive impairment (CCRI) in BC survivors may be related to the 'vascular'-toxic effects of anti-cancer therapies (Cameron et al., 2016). Indeed, both arterial stiffness and vascular function are impaired in BC patients within 15 months of initiating anti-cancer therapies (Anastasiou et al., 2023), which may be followed by neurovascular dysfunction, brain hypo- or hyper-perfusion and impaired glymphatic clearance, leading to the onset of cerebral small vessel disease and brain atrophy (Andjelkovic et al., 2023; Reeve et al., 2024).

Neurovascular units tightly regulate cerebral blood flow (CBF) to match the metabolic demands of the brain and maintain normal cognitive function (Iadecola, 2017), but damage to the neurovascular unit is associated with a reduction in CBF and the progression of and vascular-related cognitive impairment (Santisteban et al., 2023; van Dinther et al., 2024). Accordingly, resting CBF may be a clinically useful biomarker to identify patients at risk of vascular-related cognitive impairment (van Dinther et al., 2024). However, little is known about the long-term trajectory of CBF and neurovascular function in BC survivors or what interventional strategies may be effective at slowing the decline in neurovascular and neurocognitive function in BC survivors.

Regular exercise training is recognised as an effective behavioural intervention to slow or prevent the development of age-related CVD by lowering risk factors such as high blood pressure and hyperlipidaemia (Arnett et al., 2019). Higher cardiorespiratory fitness is also associated with lower dementia risk in older adults (Wang et al., 2024), which may be mediated by a reduction in cerebrovascular resistance (Smith et al., 2021) and maintenance of adequate cerebral perfusion (Tomoto et al., 2021). Furthermore, exercise training during, or shortly following chemotherapy can improve vascular function (Vear et al., 2023) and self-reported cognitive function in BC patients (Koevoets et al., 2022), However, whether exercise training incorporated into a Cardio-Oncology Rehabilitation and Exercise (CORE) programme can improve neurovascular function in long-term BC survivors is unknown. Therefore, the primary aim of this study will be to determine the effect of a CORE programme on neurovascular function in long-term breast cancer survivors.

Primary Objective:

The primary objective of this trial is to determine the effect of a CORE programme on neurovascular function in long-term breast cancer survivors.

Secondary Objective:

The secondary objective of this trial is to determine the effect of a CORE programme on neurocognitive function in long-term breast cancer survivors.

Exploratory Objective:

An exploratory objective of this study will be to determine if improvements in cardiorespiratory fitness mediate improvements in neurocognitive function in long-term breast cancer survivors.

Overall Design:

This study will be a randomised controlled trial to investigate the effect of a CORE programme on neurovascular and neurocognitive function in long-term breast cancer survivors. We will recruit n = 40 females aged 45 - 75 years old who have previously been diagnosed with stage 1 to 3 breast cancer 5 - 10 years prior to study enrolment. Participants will complete phone-based study screening and two baseline study visits to the Baker Heart and Diabetes Institute, before being randomised to a CORE programme (n = 20) or usual care (n = 20) at a 1:1 ratio. Baseline study visit one will include questionnaires, clinic blood pressure (BP), Dual-Energy X-Ray Absorptiometry (DXA) and a CPET. Participants will also be fitted with two physical activity monitors at the end of study visit one to monitor their physical activity levels over the subsequent 7 days. Baseline study visit two will include ultrasound assessments of arterial stiffness and vascular function, a neurocognitive assessment and brain MRI assessments. The 6-month CORE programme will include a 3-month exercise training programme supervised by an accredited Exercise Physiologist at the Baker Heart and Diabetes Institute, followed by 3-months of exercise training where supervision from the Exercise Physiologist is stepped-down. Exercise training adherence will be monitored throughout the step-down period by a web-based platform (Fitabase). Usual care participants will continue receiving treatment from their usual healthcare professionals. Participants will then complete two follow-up study visits following completion of the 6-month intervention period, with identical procedures to the baseline study visits. All visits and testing will occur at the Baker Heart and Diabetes Specialist Clinics, Level 4 Alfred Centre, 99 Commercial Road. All study visits will be separated by at least 24 hours.

Trial Population:

The population of interest for this trial are females living in the greater Melbourne area aged 45 - 75 years old who have previously been diagnosed with stage 1 to 3 breast cancer and have completed cardiotoxic anti-cancer therapies (e.g. anthracycline based chemotherapy or targeted radiotherapy) 5 - 10 years prior to study enrolment.

Randomisation:

Participants will then be centrally randomized to a CORE programme or usual care (see Figure 1 below) using a computerized protocol at a ratio of 1:1. Randomisation will take place at Baker Heart and Diabetes Institute and will be applied through REDCap.

Usual Care:

Participants randomised to the usual care group will be provided with their usual care by their usual healthcare professional(s). The usual care group will not be prescribed any exercise training through the study. However, they will be informed that they should aim to achieve the physical activity and exercise guidelines for Australian adults or older adults depending on their age (Care, 2024). The usual care group will not be monitored throughout the study intervention period, except for the reporting of adverse events where necessary.

Cardio-Oncology Rehabilitation and Exercise Programme:

Participants randomised to the CORE programme will receive exercise training that is analogous to cardiac rehabilitation, but Exercise Physiologists will individualise each training program using the participants baseline CPET results to maximise adherence and improve the effectiveness of the training program beyond typical cardiac rehabilitation programs. An Exercise Physiologist will supervise two training sessions a week and monitor adherence to one other independent session at home each week for the first 12 weeks of the training program whilst exercise frequency, intensity, and time is progressively increased. Supervision of the exercise training will then be stepped down gradually after 12 weeks to a fortnightly check-in to encourage intervention adherence. Patients will be provided with a training calendar and objective tools for tracking physical activity (e.g. heart rate monitor and diary). Adherence will be monitored in real-time using a research web-based platform. A similar intervention led by the PI has demonstrated excellent patient adherence (Howden et al., 2018).

Schedule of assessments

This study will involve four study visits, which will all take place at the Baker Heart and Diabetes Institute specialist clinics in the Alfred Centre. Initially, participants will be screened via telephone to assess their eligibility in the trial. Researchers will follow an approved script during telephone screening. After this initial contact, participants will be sent the PICF. Participants will then undergo the following schedule of assessments:

STUDY VISIT ONE (week -1):

Individuals will visit the testing facility after the initial eligibility assessment. Participants will be instructed to avoid caffeine for ≥ 12 hours prior to study visit 1. Furthermore, participants will be asked to avoid alcohol and strenuous physical activity for ≥ 24 hours prior to study visit 1. During study visit one, written informed consent will be obtained after the participant is comfortable with the information that they have received from the research team. After informed consent has been obtained, participants will complete questionnaires concerned with physical activity levels and menstrual cycle history. Anthropometric data will also be collected, including height, weight and body composition measured via DXA. Participants will then complete assessments of clinic blood pressure (BP), and a CPET to check their cardiorespiratory fitness. Participants will then be fitted with a hip-worn accelerometer and thigh-worn inclinometer to monitor their physical activity levels and sedentary behaviour over the subsequent seven days. Participants will also be fitted with an ambulatory blood pressure monitor (ABPM) to monitor the BP for the subsequent 24 hours.

STUDY VISIT TWO (week -1):

Participants will be instructed to fast and avoid caffeine for ≥ 12 hours prior to study visit two. Furthermore, participants will be asked to avoid alcohol and strenuous physical activity for ≥ 24 hours prior to the study visit. During study visit two, participants will complete ≥ 15 minutes of supine rest, before completing non-invasive assessments of central BP and central pulse wave velocity (cPWV) via automated Sphygmomanometry and applanation tonometry. The participant will then complete a series of duplex ultrasound scans to determine endothelium-dependent and -independent vascular function. Participants will also complete a brief neurocognitive function assessment. Participants will then complete a brain MRI protocol, compromising of 40 minutes of brain imaging whilst the participant is resting, and 8 minutes of imaging whilst the participant completes a series of 20 second breath-holds.

STUDY INTERVENTION PERIOD (weeks 1 - 26):

STUDY VISIT THREE (week 27):

Participants will complete procedures identical to those described in 'STUDY VIST ONE (week -1)'.

STUDY VISIT FOUR (week 27):

Participants will complete procedures identical to those described in 'STUDY VIST TWO (week -1)'.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 45 - 75 years old at study enrolment
* Diagnosed with stage 1 - 3 breast cancer 5 - 10 years prior to study enrolment
* Have received potentially toxic chemotherapy, including:

  * Anthracycline (any dose)
  * Trastuzumab (Herceptin) in breast-cancer with the HER2 mutation OR
  * Tyrosine kinase inhibitors (e.g. sunitinib) OR
  * Left chest radiotherapy
* ≥ 1 'traditional' CVD risk factor (I.e., Hypertension, dyslipidaemia, diabetes, obesity, smoking or family history of CVD) (Mehta et al., 2023)
* 'Physically inactive', not meeting Australian physical activity guidelines for adults or regularly participating in structured exercise training (Care, 2024).
* Eligible for Medicare
* Willing to provide written informed consent to participate in the study

Exclusion Criteria:

* Diagnosed CVD or stage B heart failure
* Diagnosed neurocognitive or cerebrovascular disease
* Diagnosed atrial fibrillation or cardiac arrythmia
* BMI ≤ 18.4 kg∙m2
* Any other contraindications to exercise testing and training that make participation in this study unsafe, determined through medical screening
* Unable to speak and understand the English language
* Contraindication to brain MRI
* Participating in another clinical research trial where randomized treatment would be unacceptable
* Oncologic (or other) life expectancy ≤ 12 months or any other medical condition (including pregnancy) that results in the belief (deemed by the Principal Investigator) that it is not appropriate for the patient to participate in this trial.

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender females.
Enrollment: 40 (Estimated)
Dates: Start 2025-11-03 (Estimated); Primary Completion 2026-07-06 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Neurovascular Function Measured via MRI-Derived Total Cerebral Blood Flow at 6 Months | 6 months
  The change in neurovascular function will be measured via total cerebral blood flow during brain magnetic resonance imaging (MRI), from pre- to post-study intervention period. Total cerebral blood flow will be measured relative to brain volume via arterial spin labeling and magnetization prepared rapid gradient echo imaging MRI scan sequences. Total cerebral blood flow will be measured in millilitres of blood per 100g of brain tissue per minute (ml.100g.min).

SECONDARY OUTCOMES:
Change from Baseline in Neurocognitive Function Measured via the Montreal Cognitive Assessment at 6 Months | 6 months
  The change in neurocognitive function will be measured via a Montreal Cognitive Assessment (MoCA) score, from pre- to post-study intervention period. The MoCA is paper-based test administered by a certified test administrator and marked on a 30-point scale (0 to 30), with lower scores indicating worse neurocognitive function.

OTHER OUTCOMES:
Determing if Changes from Baseline in Cardiorespiratory Fitness measured during Cardiopulomary Exercise Testing Mediate Improvements in Neurocognitive Function Measured via a Montreal Cognitive Assessment at 6 Months | 6 months
  Mediation analysis will be used to identify whether changes cardiorespiratory fitness - measured as maximal ventilatory intake of oxygen in millilitres per minute per kilogram of body mass (ml.min.kg) during a cardiopulmonary exercise test - from baseline to 6 months mediate improvements in neurocognitive function. Neurocognitive function will be measured via a Montreal Cognitive Assessment (MoCA) score, from pre- to post-study intervention period. The MoCA is paper-based test administered by a certified test administrator and marked on a 30-point scale (0 to 30), with lower scores indicating worse neurocognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Howden, A/Professor, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal may request access to the data from the principal investigator of the study (A/Professor Erin Howden). Proposals should be directed to erin.howden@baker.edu.au initially.
  Data requestors will also need to sign a data sharing agreement with the Baker Heart and Diabetes Institute. This contract will be reviewed by the Baker Heart and Diabetes Institute's Contracts and Compliance Manager.